CLINICAL TRIAL: NCT06862557
Title: Effects of PEMF Treatment on Patients With Mild to Moderate Dementia in a Controlled Pilot Study
Brief Title: Pulsed Electromagnetic Field Treatment With Dementia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herrick Medical LLC (Industry)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM004
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease; Lewy Body Dementia; Vascular Dementia
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Dementia, Vascular

STUDY DESIGN:
Intervention Model Description: Active treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active ECHS AD device (Experimental): Experimental intervention arm
  Interventions: Device: ECHS AD Device

INTERVENTIONS:
Device: ECHS AD Device — Pulsed electromagnetic therapy device

SUMMARY:
An open label pilot study in mild to moderate AD/ADRD patients to assess the effects of treatment with ECHS AD/ADRD pulsed electromagnetic treatment device on disease progression. Enrolled patients will receive active devices. They will treat themselves at home three times a day for 15 minutes over 120 days. Primary end point is the The Alzheimer's Disease Assessment Scale-Cognitive Subscale. Participants will be followed-up for 9 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years 2.2. Patients diagnosed with mild to moderate AD/ADRD including Alzheimer's disease, Lewy body dementia, and Vascular dementia - defined as a global CDR of 0.5 or 1 at baseline.

3. At least an eighth grade of educational achievement 4. If female, post-menopausal. 5. MMSE score between 16 and 26 (inclusive) 6. Capable of providing consent or having a surrogate (e.g., spouse, family member) capable of providing consent if participant lacks consent capacity 7. Able and willing to comply with the protocol 8. If the participant is receiving a cholinesterase inhibitor and/or memantine, such medication has been prescribed for at least 3 months prior to screening and the dose is stable for at least 60 days prior to screening (that dose needs to be maintained throughout the period of this study) 10. Physical clearance for study participation as evaluated by the clinician

Exclusion Criteria:

1. The patient lacks capacity to consent to study participation and no surrogate is available to provide consent
2. The patient does not have a study partner who would be available for interview
3. History of epileptic seizures or epilepsy
4. Has Frontotemporal Dementia
5. Currently taking medication that lowers the seizure threshold, excluding blood thinners
6. Is currently taking anti-amyloid monoclonal antibodies (past treatment is allowed if termination of treatment occurred at least 3 months prior to the baseline visit).
7. Presence of depression, bipolar disorder, a psychotic disorder, or any other neurological or psychiatric condition (whether now or in the past), which the Investigator finds as interfering with the study
8. Severe agitation that would interfere with study procedures
9. Alcoholism or substance use disorder as defined by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) within last 5 years (addicted more than one year and or in remission less than 3 years) or severe sleep deprivation
10. Major surgery (defined as any major abdominal, vascular or thoracic surgery requiring general anesthesia and resulting in a period of >1 week hospitalization) within 4 weeks
11. Head anatomy that interferes with the fit of the treatment device
12. Participation in another clinical trial within the previous 30 days
13. Metal implants in the head, (i.e., cochlear implants, implanted brain stimulators and neurostimulators, aneurysm clips) with the exception of metal implants in mouth
14. Criteria to exclude participants from the blood draw study:

Any condition that may significantly increase risks associated with blood draws

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) | Change between day 0, and 45, 90, 135, 180 days
  Assessment consisting of 11 tasks, taking up to 30mins, to measure the severity of cognitive dementia symptoms. Score 0-70, Higher number, more severity.

SECONDARY OUTCOMES:
Mini-Mental Status Exam (MMSE) | Change between day 0, and 45, 90, 135, 180 days
  Clinician assessment of cognitive impairment. Scoring 0-30, lower score, more severity
Quality of Life Scale | Change between day 0, and 45, 90, 135, 180 days
  Clinician assessment of cognitive impairment. Scored 0-7, higher score, greater severity
Global Deterioration questionnaire | Change between day 0, and 45, 90, 135, 180 days
  Clinician assessment of cognitive impairment. Scored 0-7, higher score, greater severity
Side-Effects Questionnaire | Change between day 0, and 45, 90, 135, 180 days
  Self-report of side-effects
Clinical Dementia Rating (CDR) sum of boxes (CDR-SB) | Change between day 0, and 90, 180 days
  CDR-SB assesses the severity and progression of dementia

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided